CLINICAL TRIAL: NCT06504576
Title: Effect of Cilostazol in Promoting Hematoma Clearance After Intracerebral Hemorrhage: A Phase-II Open Label Study
Brief Title: Effect of Cilostazol in Promoting Hematoma Clearance After Intracerebral Hemorrhage
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202311026MINC
Record Dates: First submitted 2024-03-25; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-01

CONDITIONS: ICH - Intracerebral Hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage | interventions — Cilostazol; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cilostazol treatment with conventional treatment (Experimental): The drug treatment group will receive two consecutive weeks of Cilostazol two days after admission and receive conventional treatment as well.
  Interventions: Drug: Cilostazol 50 MG Oral Tablet
- Conventional treatment only (Placebo Comparator): The conventional treatment group will receive conventional internal medicine treatment only.
  Interventions: Procedure: Conventional internal medicine treatment

INTERVENTIONS:
Drug: Cilostazol 50 MG Oral Tablet — Two consecutive weeks of Cilostazol (50mg BID) two days after admission
  Other Names: Pletal 50 MG Oral Tablet
  Arms: Cilostazol treatment with conventional treatment
Procedure: Conventional internal medicine treatment — Receives only conventional internal medicine treatment
  Arms: Conventional treatment only

SUMMARY:
Intracerebral hemorrhage (ICH) is a dangerous form of stroke with high mortality rate. Other than evacuating the hematoma with surgical procedures, there is no current effective internal medicine treatment. Currently, there are many novel internal medicine treatment under development, one of which is the promotion of endogenous hematoma clearance. Our team recently found out that the meningeal lymphatic system plays an important role in clearing hematoma post-ICH, meaning that promoting the drainage function of the meningeal lymphatic system may have a certain level of help for improving the prognosis of ICH.

Cilostazol is an anti-PDE3 type antiplatelet agent with the function of preventing peripheral arterial occlusion disease and stroke. Cilostazol has been proven to promote lymphatic endothelial cell proliferation and the drainage function of the lymphatic system. Our animal research points out that Cilostazol speeds up hematoma clearance post-ICH and generates neuroprotective effects, thereby improving prognosis and providing a new internal medicine treatment for ICH.

Due to the fact that there is no clinical trial looking into the hematoma resorption effect of Cilostazol in ICH patients, this trials aims to understand the safety and hematoma resorption efficacy of Cilostazol in acute ICH patients. Investigators estimate to enroll 100 patients in National Taiwan University Hospital (NTUH) within 3 years. The patients would be randomized into two groups, one receiving Cilostazol (two weeks, 50mg BID) and conventional treatment, and the other group receiving only conventional treatment. Investigators will assess the patients' neurological outcome and functional aspects (NIHSS, modified Rankin Scale) two weeks / one month / three months after ICH. Investigators will also use MRI to measure hematoma size to evaluate hematoma resorption (primary endpoint and safety endpoint). MRI will also be used to measure the drainage effect of the meningeal lymphatics.

DETAILED DESCRIPTION:
After the subject is sent to the emergency department, he/she will receive a CT scan to evaluate the size and location of the hematoma. ICH score will be used to evaluate the severity of the subject. The subject will then be randomized to the drug treatment group or the conventional treatment group. The drug treatment group would receive two consecutive weeks of Cilostazol (50mg BID) two days after admission and conventional treatment, whereas the conventional treatment group only receives conventional internal medicine treatment. The subject would receive an MRI scan after finishing his/her course of Cilostazol (16 +/- 2 days post-ICH) to assess the size of the hematoma and brain meningeal lymphatic drainage effects. Investigators will gather information from the subject such as age, sex, vascular risk factors, past antithrombotic treatment history and past stroke history. Basic biochemistry panels (including coagulation function and complete blood count) and clinical data (including neurological deficits and blood pressure on admission) will also be gathered. Investigators are scheduled to perform the NIHSS scale and the modified Rankin Scale 1/14/30/90 days after ICH to evaluate the level of disability.

ELIGIBILITY:
Inclusion criteria:

1. Adult patients (at least 20 years old, no upper limit)
2. ICH located in the thalamus or basal ganglia.
3. ICH score less than 3 (hematoma volume no greater than 15 ml) and was admitted within 24 hours since onset.
4. The patient or his/her legal representative agrees to join this trial and accept the arrangements of tests within this trial.

Exclusion criteria:

1. ICH in the cerebral lobar areas or under the cerebellar tentorium, or ICH score greater than 3.
2. Surgical intervention was suggested after evaluation
3. Subject has brain trauma, structural brain disease, metabolic brain disease, neuroinflammatory disease and brain tumor.
4. Subject that cannot accept image examination, including but not limited to unable to cooperate, disruption of image quality due to agitation, unstable hemodynamics, has MRI-incompatible pacemakers, has aneurysmal clip or claustrophobia.
5. Subject has contraindication for using contrast medium, including chronic kidney failure (CCr < 30ml/min) or allergic to contrast medium.
6. Subject is currently pregnant or is scheduled to be pregnant within the following 6 months.
7. Subject is taking other antithrombotics, including antiplatelet drugs (Aspirin, Clopidogrel, Ticagrelor) and oral anticoagulative (Warfarin, Dabigatran, Rivaroxaban Apixaban, Edoxaban) when ICH happened.
8. Subject has contraindication to using Cilostazol, such as heart failure of any severity, coagulative disorders, ventricular tachycardia, ventricular fibrillation, multi-focal ventricular arrhythmia, severe tachycardic arrhythmia, unstable angina, myocardial infarction in recent 6 months, or had received coronary intervention.
9. Life expectancy less than 3 months.
10. Subject has known allergy to drugs used in the trial and was designated not suitable to enroll in this trial by the host.
11. Subject or his/her legal representative does not agree to join this trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome | 16 days post-ICH
  Hematoma size comparison at 16 days post-ICH in the drug treatment group and conventional treatment group by measuring MRI T2WI. Whether taking two consecutive weeks of Cilostazol causes hematoma expansion.

SECONDARY OUTCOMES:
Secondary outcome 1 | 16/30/90 days post-ICH
  Subject's National Institute of Health Stroke Scale (0-42) score change 16/30/90 days post-ICH.
  With higher scores indicating greater severity
Secondary outcome 2 | 30/90 days post-ICH
  Subject's mRankin Scale score(0-6) change 30/90 days post-ICH compared with pre-treatment status. (the ratio of mRS score 0-1 and 0-2, with higher scores indicating greater severity.)
Secondary outcome 3 | 16 days post-ICH
  The difference of DCE-MRI time to maximal intensity between drug treatment group and conventional treatment group.
Secondary outcome 4 | 16 days post-ICH
  Hematoma resorption rate difference between drug treatment group and conventional treatment group 16 days post-ICH.

OTHER OUTCOMES:
Safety outcome 1 | 90 days
  Patient develops hematoma expansion
Safety outcome 2 | Within 16 days
  Patient requires surgical evacuation of hematoma or open craniotomy for pressure relief
Safety outcome 3 | Within 16 days
  Any adverse event or severe adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-Hsi Tsai, MD, PhD, Principal Investigator — Department of Neurology, National Taiwan University Hospital

IPD SHARING:
Plan to Share IPD: No